CLINICAL TRIAL: NCT03757442
Title: An Observational Study of the Association Between the Perioperatively Measured Peripheral Perfusion Index, Postoperative Complications and Mortality in Acute Surgical Patients
Brief Title: Peripheral Perfusion Index in Acute Surgical Patients
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Agerskov, MD, Research Fellow, Hvidovre University Hospital
Other Study IDs: W217038300-2018-77
Record Dates: First submitted 2018-10-15; First posted 2018-11-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2019-10

CONDITIONS: Fracture of Hip; Ileus; Perforated Viscus; Anastomotic Leak
MeSH Terms: conditions — Hip Fractures; Ileus; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction Perioperative haemodynamic instability is associated with postoperative morbidity and mortality. Macrocirculatory parameters, such as the conventionally obtained mean arterial blood pressure and cardiac output, may be uncoupled from the microcirculation during sepsis and severe blood loss and may not necessarily be optimal resuscitation parameters. The peripheral perfusion index (PPI) is derived from the pulse oximetry signal and reflects perfusion. Reduced peripheral perfusion is associated with morbidity in critically ill patients and in patients following acute surgery. We hypothesize that patients with low intraoperative PPI demonstrate high frequency of postoperative complications and mortality regardless of blood pressure.

Methods and analysis We plan to conduct a prospective observational cohort study in patients undergoing acute non-cardiac surgery (November 1st, 2017 to October 31st, 2018) at two University Hospitals. Data will be collected prospectively from patient records including patient demographics, comorbidity and intraoperative hemodynamic values, with PPI as the primary exposure variable, and postoperative complications and mortality within 30 and 90 days as outcome variables. We primarily assess association between PPI and outcome in multivariate regression models. Secondly, the predictive value of PPI for outcome, using area under the receiver operating characteristics curve is assessed.

Ethics and dissemination Data will be reported according to The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE). Results will be published in a peer reviewed journal. The study is approved by the regional research ethics committee, storage and management of data has been approved by the Regional Data Protection Agency, and access to medical records is approved by the hospital board of directors at the involved hospitals and departments.

DETAILED DESCRIPTION:
Background Perioperative haemodynamic instability is associated with postoperative morbidity and mortality. Patients undergoing acute major abdominal or hip fracture surgery have high complication rates and account for a major part of overall postoperative mortality in developed countries. These patients are often frail, with multiple comorbidities making them vulnerable to anaesthesia and surgery. Despite the benefit of a multidisciplinary effort to improve perioperative care, such patients demonstrate a high risk of complications and death. Conventional perioperative haemodynamic monitoring is often based only on heart rate (HR) and mean blood pressure (MAP). Although perioperative hypotension is associated with complications in major surgery, blood pressure is often an inadequate marker of perioperative organ perfusion, consequently leading to little precision in administration of fluid and vasoactive medication. Minimally-invasive haemodynamic monitoring of cardiac output (CO), and goal directed therapy based on stroke volume optimization, has been associated with improved outcome in major elective surgery, but high quality evidence for the advantage of such monitoring in emergency surgery is sparse.

Macrocirculatory parameters such as MAP and CO may be uncoupled from the microcirculation during sepsis and severe blood loss due to sympathetic or medically induced vasoconstriction, and as such, these parameters are not necessarily optimal for resuscitation.

Assuming that blood flow is directed from peripheral tissue to vital organs during progressive stages of circulatory impairment and shock, a non-invasive method to detect impaired peripheral perfusion could be a relevant endpoint.

The peripheral perfusion index (PPI) has the advantage that is derived from the photoelectric plethysmographic pulse oximetry signal most likely obtained in all patients for evaluation of arterial oxygen saturation (SAT) already in the emergency room and continued during and after surgery as in wards and in the ICU. The PPI reflects the ratio between the pulsatile and non-pulsatile component of the arterial waveform as assessed by light traversing the tissue addressed, most often the finger, and it decreases in response to hypoperfusion.Thus, PPI reflects changes in peripheral perfusion and blood volume and reduced peripheral perfusion is associated with morbidity following acute surgery, in critically ill patients, and patients presenting septic shock. However, it remains uncertain which threshold for PPI should trigger intervention in patients undergoing acute surgery reflecting that evaluation is made only in relatively small populations of mixed medical and surgical patients.

Hypothesis We hypothesize that PPI reflects impaired peripheral circulation and that patients with low intraoperative PPI, independent of MAP, have higher risk of postoperative complications and mortality than patients with normal or high PPI.

Objectives The main objective of this study is to evaluate the association between intraoperative PPI and outcome defined as severe postoperative complications and 30- and 90-days mortality. Secondly, we assess the predictive value of intraoperative PPI in relation to outcome and evaluate whether PPI has better prediction of adverse outcome than the commonly used MAP thresholds and try to establish intervention thresholds for PPI that in acute non-cardiac surgical patients.

ELIGIBILITY:
Inclusion Criteria:

Orthopedic surgery patients with fracture of the hip booked for or having performed procedures with the following procedural codes: KNFB02, KNFJ81, KNFJ51, KNFJ52, KNFJ70 representing arthroplasty, intra-medullar nailing, and screws respectively.

For abdominal surgery patients we include patients booked for acute laparoscopy for diagnostic purposes (KJAH01) and explorative laparotomy (KJAH00). To identify all patients having performed acute abdominal surgery, we also include surgery related to ileus: KJFK00, KJFK01, KJFK10, KJAP00, KJAP01, KJFK96, KJFK97, any perforation of vicera: KJDA60, KJDA70, KJDA80, and any ischemic condition of the gut: KJFB00, KJFB01, KJFB33, KJFB34, KJFB96, KJFB97.

Exclusion Criteria:

* No sampling of PPI registered
* Foreign/temporary civil registration number that prevents follow up
* Earlier enrollment in cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years of age having performed acute abdominal or orthopedic surgery from 1th November 2017 through 31th October 2018 at Hvidovre and Bispebjerg University Hospitals. Study subjects will be obtained from the hospitals electronic medical records via specific procedural- or diagnostic codes representing the acute orthopedic or abdominal surgery in the specified one-year period.
Sampling Method: Probability Sample
Enrollment: 1338 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Any severe complication or death | 30 days
  Severe postoperative complications (Clavien Dindo III-IV) or death (Clavien Dindo V)

SECONDARY OUTCOMES:
Any severe complication or death | 90 days
  Severe postoperative complications (Clavien Dindo III-IV) or death (Clavien Dindo V)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agerskov M, Thusholdt ANW, Hojlund J, Meyhoff CS, Sorensen H, Wiberg S, Secher NH, Bang Foss N. Protocol for a multicentre retrospective observational cohort study in Denmark: association between the intraoperative peripheral perfusion index and postoperative morbidity and mortality in acute non-cardiac surgical patients. BMJ Open. 2019 Nov 21;9(11):e031249. doi: 10.1136/bmjopen-2019-031249. PMID 31753878